CLINICAL TRIAL: NCT05965674
Title: The Effect of Sacral Erector Spinae Plane Block on Post-Hemorrhoidectomy Pain
Brief Title: Sacral Erector Spinae Plane Block Effect on Post-Hemorrhoidectomy Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Aydın Mermer, Anesthesiologist, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KonyaCityH Study Hemo
Record Dates: First submitted 2023-07-04; First posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain
Keywords: Sacral Erector Spinae Plane Block; Post-Hemorrhoidectomy Pain; Analgesic consumption
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The sacral ESPB group (Group S) (Active Comparator): Patients in Group S underwent a procedure where a high-frequency linear ultrasound probe (Clarius, 205-2980 Virtual Way, Vancouver, BC, Canada V5M 4X3 MyLabFive; Esaote Europe BV Philipsweg 1 6227 AJ, Maastricht, the Netherlands) was positioned on the transverse plane, specifically on the fifth spinous process. The probe was then moved downwards to visualize the first and second median sacral crest. Next, the transducer was placed 3-4 cm laterally to the second medial sacral crest in order to visualize the intermediate sacral crest. In the interfascial plane, a total of 20 mL of local anesthetic solution (comprised of 10 mL bupivacaine 0.5%, 5 mL lidocaine 2%, and 5 mL normal saline) was injected between the erector spinae muscles and the intermediate sacral crest. The same procedure was performed on the contralateral side.
  Interventions: Procedure: Sacral Erector Spinae Plane Block
- The control group (Group N) (No Intervention): It will not be performed any extra intervention, just rutin clinic protocol.

INTERVENTIONS:
Procedure: Sacral Erector Spinae Plane Block — The transducer will be placed 3-4 cm laterally to the second medial sacral crest in order to visualize the intermediate sacral crest. In the interfascial plane, a total of 20 mL of local anesthetic solution (comprised of 10 mL bupivacaine 0.5%, 5 mL lidocaine 2%, and 5 mL normal saline) will be injected between the erector spinae muscles and the intermediate sacral crest. The same procedure will be performed on the contralateral side.
  Arms: The sacral ESPB group (Group S)

SUMMARY:
Hemorrhoids are commonly observed surgical conditions affecting the anorectal area, characterized by symptoms such as pain, bleeding, and the presence of a protruding mass from the anal opening. Fear of postoperative pain is one of the most important factors for patients to avoid surgical interventions. Postoperative pain is a significant concern, with over 80% of patients encountering moderate to severe pain.

The main aim is to evaluate ESPB from the sacral level would result in effective analgesia following hemorrhoidectomy. It is also aimed if sacral ESPB would reduce the use of additional analgesics after hemorrhoidectomy and increase patient satisfaction. In this prospective, randomized, controlled trial, our main objective was to examine the postoperative analgesic effects of sacral ESPB following hemorrhoidectomy.

DETAILED DESCRIPTION:
Hemorrhoids are commonly observed surgical conditions affecting the anorectal area, characterized by symptoms such as pain, bleeding, and the presence of a protruding mass from the anal opening. Fear of postoperative pain is one of the most important factors for patients to avoid surgical interventions. Postoperative pain is a significant concern, with over 80% of patients encountering moderate to severe pain. This heightened pain level contributes to an elevated risk of complications including atelectasis, thromboembolism, myocardial ischemia, cardiac arrhythmia, electrolyte imbalance, urinary retention, and ileus. The two main unresolved issues following surgery are postoperative pain and urinary retention. In addition to improving patient satisfaction, pain management will decrease urinary retention and constipation, especially in the first 24 hours following surgery. According to earlier research, even with analgesic therapy, 20% to 40% of patients who underwent hemorrhoidectomy would experience severe postoperative pain. Commonly used pain relievers like nonsteroidal anti-inflammatory drugs, paracetamol, and opioids often come with adverse effects such as dizziness, nausea, vomiting, and constipation and can even lead to tolerance. These side effects could prevent a full recovery and result in a poor prognosis. Bilateral pudendal nerve blocks are said to significantly reduce postoperative pain, but they are technically difficult and require specific positioning. Furthermore, the administration of pudendal nerve block carries the risk of potential complications, including hematoma formation, sciatic nerve injury, and accidental rectal puncture. Therefore, an alternative analgesic method with minimal adverse effects would be beneficial.

The erector spinae plane block (ESPB) was initially introduced as an interfascial plane block performed at the upper thoracic levels with the purpose of alleviating neuropathic pain. Subsequently, its application expanded to encompass a range of thoracic interventions, including mastectomy, video-assisted thoracoscopy (VATS), and cardiac surgery, while also being utilized at lumbar levels for procedures such as abdominal surgery, prostatectomy, lumbar spine surgery, total hip arthroplasty, and proximal femur surgery. A newly introduced method called the sacral Erector Spinae Plane Block (ESPB) has been recently documented in scientific literature. Case studies have demonstrated its effectiveness in various surgical procedures. Specifically, it has shown promise in managing radicular pain at the L5-S1 level after sex reassignment surgery and hypospadias surgery, as well as providing analgesia for the posterior branches of the sacral nerves during pilonidal sinus surgery.

The main hypothesis is that performing ESPB from the sacral level would result in effective analgesia following hemorrhoidectomy. It is also hypothesized that sacral ESPB would reduce the use of additional analgesics after hemorrhoidectomy and increase patient satisfaction. In this prospective, randomized, controlled trial, the main objective is to examine the postoperative analgesic effects of sacral ESPB following hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

* being between the ages of 18 and 65,
* having an ASA status of 1-2.

Exclusion Criteria:

* under the age of 18, pregnant individuals,
* significant hematopoietic, cardiovascular, liver, or kidney disorders,
* patients unable to comply with medical instructions, individuals on anticoagulant therapy, and those with contraindications to regional anesthetic agents or a history of previous hemorrhoidectomy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
pain intensity at rest and in motion evaluated with an NRS (0-10, 0 = no pain, 10 = worst pain) at 0, 2, 4, 6, 12, and 24h. | Perioperative period
  The primary outcome is pain score at rest and in motion evaluated with an NRS (0-10, 0 = no pain, 10 = worst pain) at 0, 2, 4, 6, 12, and 24h.

SECONDARY OUTCOMES:
The cumulative doses of tramadol, the number of patients who required rescue medication postoperatively, and QoR-15T patient recovery quality. | Perioperative period
  The secondary outcome measures are the cumulative doses of tramadol, the number of patients who required rescue medication postoperatively, and QoR-15T patient recovery quality.

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Mermer, Konya, Selcuklu, Turkey (Türkiye)